CLINICAL TRIAL: NCT07154654
Title: Prospective, Long Term, Observational Study (Patient Registry) of Paediatric Myotonic Disorders From Birth to Less Than Six Years of Age Who Are Treated With Mexiletine (PEGASUS Study).
Brief Title: Prospective, Long Term, Observational Study (Patient Registry) of Paediatric Myotonic Disorders
Status: Recruiting | Type: Observational
Sponsor: Lupin Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: MEX-NM-401
Record Dates: First submitted 2025-07-24; First posted 2025-09-04 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Myotonic Disorders
MeSH Terms: conditions — Myotonic Disorders | interventions — Mexiletine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Infants and children aged between 6 months to less than 6 years.
  Interventions: Drug: Mexiletine
- Cohort 2: Neonates and infants from birth to less than 6 months.
  Interventions: Drug: Mexiletine

INTERVENTIONS:
Drug: Mexiletine — Non interventional

SUMMARY:
This is a prospective, open-label, multi-centre, single arm, registry study to collect standard relevant clinical and epidemiological data during routine medical evaluation and treatment in paediatric patients with myotonic disorders who are being treated with mexiletine therapy according to the physician.

DETAILED DESCRIPTION:
This is a prospective, open-label, multi-centre, single arm, registry study to collect standard relevant clinical and epidemiological data during routine medical evaluation and treatment in paediatric patients with myotonic disorders who are being treated with mexiletine therapy according to the physician.

Patients who meet the eligibility criteria will be enrolled in 2 cohorts by age groups although cohorts are not enrolled sequentially (cohort definition is to assure minimum requirements for meeting PIP agreements).

Cohort 1 - Infants and children aged between 6 months to less than 6 years. Cohort 2 - Neonates and infants from birth to less than 6 months. The overall treatment duration follow-up for each cohort will be at least 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients from birth to less than 6 years
2. A genetically confirmed diagnosis of NDM or DM (DM1or DM2), as per the treating clinician.
3. Presence of clinical symptoms of myotonia (hand grip myotonia, myotonia in the leg muscles, any other myotonia symptoms) to be confirmed by the treating clinician.
4. Patients already receiving mexiletine treatment or who are clinically considered for mexiletine treatment as per the treating physician judgement.
5. No history of or significant cardiac abnormalities as determined by a cardiologist's assessment of the ECG and echocardiogram performed prior to enrolment in the study or as per the treating physician standard of care (NaMuscla SmPC, 2023)
6. No known history or signs and symptoms of any significant liver disorder as per treating physician.
7. No known clinically relevant abnormal laboratory investigations for haematology, biochemistry, and urinalysis values at screening (or based on values obtained within 3 months prior to screening in patient's medical record) that could affect the study objectives as judged by the treating physician.
8. Parent or legal guardian able to provide consent/assent to study participation and to sign the written informed consent or non-opposition as per local regulatory requirements prior to study entry and perform any study-related activity. -

Exclusion Criteria:

1. Any contraindication to mexiletine as listed in the Namuscla Summary of Product Characteristics (SmPC) (NaMuscla SmPC, 2023)

   1. Hypersensitivity to the active substance, or to any of the excipients
   2. Hypersensitivity to any local anaesthetic
   3. Ventricular tachyarrhythmia
   4. Complete heart block (i.e., third-degree atrioventricular block) or any heart block susceptible to evolve to complete heart block (first-degree atrioventricular block with markedly prolonged PR interval (≥ 200 ms) and/or wide QRS complex (≥ 120 ms), second-degree atrioventricular block, bundle branch block, bifascicular and trifascicular block),
   5. QT interval > 450ms
   6. Myocardial infarction (acute or past), or abnormal Q-waves
   7. Symptomatic coronary artery disease
   8. Heart failure with ejection fraction <50%
   9. Atrial tachyarrhythmia, fibrillation or flutter
   10. Sinus node dysfunction (including sinus rate < 50 bpm)
   11. Co-administration with medicinal products inducing torsades de pointes.
   12. Co-administration with medicinal products with narrow therapeutic index
2. Any other neurological or psychiatric condition that might affect the study assessments, as per the treating clinician.
3. Any clinically significant illness, laboratory findings, ECG, or other clinical symptoms, which in the opinion of the treating physician could affect the patient's optimal participation in the study
4. Receiving strong inducers or inhibitors of CYP2D6 or CYP1A2 or planned to receive them, during the subject participation (See section 4.1.5.1 Prohibited medications).
5. Any concurrent illness, or medications which could affect the muscle function, and confound the results according to the treating physician.
6. Seizure disorder, diabetes mellitus requiring treatment by insulin.

Max Age: 6 Years | Sex: All
Age Groups: Child
Study Population: The study population will include male and female children from birth to less than 6 years of age with clinical symptoms or signs of myotonic disorders, normal electrocardiogram (ECG) exam and genetic confirmation of the diagnosis i.e., non-dystrophic myotonia (NDM), or myotonic dystrophy (DM) type 1 (DM1), or DM type 2 (DM2), and who comply with the inclusion / exclusion criteria.
  Patients will be enrolled consecutively at each site in order to minimize selection bias
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2027-11-22 (Estimated); Study Completion 2028-02-22 (Estimated)

PRIMARY OUTCOMES:
To assess long-term safety by collection of SAEs, AEs, AESIs, changes in frequency, treatment interruptions | Baseline to 24 months
  Number and frequency of adverse events (AEs), serious adverse events (SAEs) and AE leading to treatment discontinuation, throughout the study while on treatment with mexiletine; Incidence of adverse events of special interest (AESI), namely: Severe Cutaneous Adverse Reactions (SCARs) & Cardiac arrhythmia. Increased frequency of seizure episodes in patients with epilepsy; Any changes in frequency, treatment interruptions of mexiletine

SECONDARY OUTCOMES:
To assess the suitability of mexiletine administration | Baseline to 24 months
  To assess the suitability of mexiletine administration using available formulations including, where appropriate, capsules or opening and sprinkling contents in food or drink according to the child´s age (from birth to less than 6 years) and ability to swallow.
To understand how mexiletine is used by clinicians | Baseline to 24 months
  To understand how mexiletine is used by clinicians who have previously decided to use mexiletine for the treatment of myotonia in myotonic disorder patients, from birth to less than 6 years over a at least 2 years period, to establish risk:benefit conclusions.
Description over time of outcomes of mexiletine use | Baseline to 24 months
  Description over time of outcomes of mexiletine use including dosing, formulation used, method of administration, acceptability and palatability as per the data collected by the treating physician according to age and cohort.
The treating physician with elaborate a brief text with risk-benefit conclusions | Baseline to 24 months
  Description over time of any efficacy outcomes obtained from clinically indicated tests as per the treating physician typical clinical practice and according to patient's age and cohort.

OTHER OUTCOMES:
Description over time of any efficacy outcomes | Baseline to 24 months
  Description over time of any efficacy outcomes obtained from clinically indicated tests as per the treating physician typical clinical practice and according to patient's age and cohort.
Clinical Global Impression (CGI) Scores | Baseline to 24 months
  Clinical Global Impression (CGI) Scores given to caregivers and assessed by the investigators. Efficacy will be evaluated on a 4-point scale as very efficient, good, fair or poor.

CONTACTS AND LOCATIONS:
Overall Officials: Catharine Sarret, MD, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Centre Hospitalier Universitaire de Clermont-Ferrand, Clermont-Ferrand, France